CLINICAL TRIAL: NCT06923930
Title: Impact of a Cueing Device on Upper Extremity Muscle Strength in Swimmers: A 6-Week Training Protocol Using Scapular Stabilization Exercises.
Brief Title: Impact of a Cueing Device on Upper Extremity Muscle Strength in Swimmers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, Kevin Strehler, Assistant Professor of Physical Therapy, University of South Alabama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2305310-1/2304240-1
Record Dates: First submitted 2025-03-29; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers Only
Keywords: External cue; Shoulder Stability; Strength Exercise; Adolescent Swimmer
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise Program Alone Exercise Program with External Cueing Device
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shoulder Stabilization Exercise (Active Comparator): Protocol contains 8 exercises ("I", "Y", "T", "i", "w", alternating arm "I"/"i", "n", and supine serratus punch) completed for 8 repetitions each for 3 weeks, and in weeks 4-6 completed at 2 sets of 8 repetitions each. Standard group coaching assistance will be provided.
  Interventions: Other: Exercise
- Shoulder Stabilization Exercise with External Cueing Device (Experimental): Protocol contains 8 exercises ("I", "Y", "T", "i", "w", alternating arm "I"/"i", "n", and supine serratus punch) completed for 8 repetitions each for 3 weeks, and in weeks 4-6 completed at 2 sets of 8 repetitions each. External cueing device provides movement pattern constraint and an external target zone for the individual for each exercise. Standard group coaching assistance will be provided.
  Interventions: Device: External Cueing Device; Other: Exercise

INTERVENTIONS:
Device: External Cueing Device — A portable product that provides movement pattern constraints to ensure improved exercise form, and provides a target zone for exercise effort
  Arms: Shoulder Stabilization Exercise with External Cueing Device
Other: Exercise — Shoulder stabilization exercise protocol contains 8 exercises ("I", "Y", "T", "i", "w", alternating arm "I"/"i", "n", and supine serratus punch) completed for 8 repetitions each for 3 weeks, and in weeks 4-6 completed at 2 sets of 8 repetitions each.

SUMMARY:
The goal of this study is to find out if a tool called an external cueing device (ECD) can help young swimmers improve their shoulder function. An ECD is a tool that limits arm movement and gives the swimmer a target to focus on while doing exercises. The main questions this study will answer are:

* Does using an ECD during certain exercises improve muscle strength?
* Does using an ECD while exercising help with shoulder stability?

Participants will:

* Test their shoulder muscle strength and stability at the beginning of the study.
* Complete 8 exercises as part of their regular dry-land training program for 6 weeks.
* Repeat the same tests after 3 weeks and again at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer Adolescent Swimmers
* Member of CMSA

Exclusion Criteria:

* Swimmers under the age of 11 years of age.
* Swimmers that are not registered as athletes through United States Swimming.
* Swimmers that are not enrolled in Age Group III, Senior 1, Senior 2, or Senior 3
* Swimmers not attending practice due to an injury (i.e., shoulder, back, etc.).
* Swimmers currently not participating in a dryland program offered through CMSA.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in isometric muscle torque production at 180 degrees shoulder abduction | Baseline, 3 weeks, 6 weeks.
  Handheld dynamometer assessment of force production times lever arm distance (Newton.meters) of prone shoulder elevation in 180 degrees of abduction completed at baseline, after 3 and 6 weeks of the training program.
Change from baseline in isometric muscle torque production at 135 degrees shoulder abduction | Baseline, 3 weeks, 6 weeks.
  Handheld dynamometer assessment of force production times lever arm distance (Newton.meters) of prone shoulder elevation in 135 degrees of abduction completed at baseline, after 3 and 6 weeks of the training program.
Change from baseline in isometric muscle torque production at 90 degrees shoulder abduction | Baseline, 3 weeks, 6 weeks.
  Handheld dynamometer assessment of force production times lever arm distance (Newton.meters) of prone shoulder elevation in 90 degrees of abduction completed at baseline, after 3 and 6 weeks of the training program.
Change from baseline in modified Athletic Shoulder Test at 180 degrees shoulder abduction | Baseline, 3 weeks, 6 weeks.
  Maximum isometric force production with lying prone into a handheld dynamometer at a given lever arm distance results in muscle torque (Newton.meters) reading. This portion of the test is conducted at 180 degrees of abduction.
Change from baseline in modified Athletic Shoulder Test at 135 degrees shoulder abduction | Baseline, 3 weeks, 6 weeks.
  Maximum isometric force production with lying prone into a handheld dynamometer at a given lever arm distance results in muscle torque (Newton.meters) reading. This portion of the test is conducted at 135 degrees of abduction.
Change from baseline in modified Athletic Shoulder Test at 90 degrees shoulder abduction | Baseline, 3 weeks, 6 weeks.
  Maximum isometric force production with lying prone into a handheld dynamometer at a given lever arm distance results in muscle torque (Newton.meters) reading. This portion of the test is conducted at 90 degrees of abduction.
Closed Kinetic Chain Upper Extremity Stability Test Power Score | Baseline, 6 weeks.
  Two strips of tape are placed 36 inches apart. Participants assume a push up position (male) or pushup on knees (Female) and are instructed to reach across and touch the opposing hand alternating arms. Maximum number of touches in 15 seconds is recorded. Normalization is made by multiplying the raw touch score by 0.68 x Subject weight in Kg (representing the mass on the head arms and trunk) and dividing by the 15 seconds. Higher number indicates increased shoulder stability.

SECONDARY OUTCOMES:
Closed Kinetic Chain Upper Extremity Stability Test Raw Touch Score | Baseline, 6 weeks.
  Two strips of tape are placed 36 inches apart. Participants assume a push up position (male) or pushup on knees (Female) and are instructed to reach across and touch the opposing hand alternating arms. Maximum number of touches in 15 seconds is recorded. Higher number of touches indicates increased shoulder stability
Closed Kinetic Chain Upper Extremity Stability Test Touch Score | Baseline, 6 weeks.
  Two strips of tape are placed 36 inches apart. Participants assume a push up position (male) or pushup on knees (Female) and are instructed to reach across and touch the opposing hand alternating arms. Maximum number of touches in 15 seconds is recorded. Touches are adjusted for subject height by dividing raw touch by subject height (in inches based on prior literature). Higher number of touches indicates increased shoulder stability
Maximal Prone Arm Elevation at 180 degrees abduction | Baseline, 3 weeks, 6 weeks.
  Distance from floor to wrist crease, measured in cm.
Maximal Prone Arm Elevation at 135 degrees abduction | Baseline, 3 weeks, 6 weeks.
  Distance from floor to wrist crease, measured in cm.
Maximal Prone Arm Elevation at 90 degrees abduction | Baseline, 3 weeks, 6 weeks.
  Distance from floor to wrist crease, measured in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Fredericka G. Evans Cultural Centre, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Oliveira VM, Pitangui AC, Nascimento VY, da Silva HA, Dos Passos MH, de Araujo RC. TEST-RETEST RELIABILITY OF THE CLOSED KINETIC CHAIN UPPER EXTREMITY STABILITY TEST (CKCUEST) IN ADOLESCENTS: RELIABILITY OF CKCUEST IN ADOLESCENTS. Int J Sports Phys Ther. 2017 Feb;12(1):125-132. PMID 28217423
- [Background] Tooth C, Forthomme B, Croisier JL, Gofflot A, Bornheim S, Schwartz C. The Modified-Athletic Shoulder Test: Reliability and validity of a new on-field assessment tool. Phys Ther Sport. 2022 Nov;58:8-15. doi: 10.1016/j.ptsp.2022.08.003. Epub 2022 Aug 30. PMID 36088802